CLINICAL TRIAL: NCT06428578
Title: Enhancing Food as Medicine Interventions for Food Insecure Postpartum Women in Central Texas
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Texas Health Science Center, Houston (Other)
Collaborators: American Heart Association (Other)
Responsible Party: Principal Investigator, Alexandra van den Berg, Professor, The University of Texas Health Science Center, Houston
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HSC-SPH-23-0795; 24FIM1264463 (Other Grant/Funding Number: American Heart Association)
Record Dates: First submitted 2024-05-20; First posted 2024-05-24 (Actual); Last update posted 2024-05-24 (Actual); Status verified 2024-05

CONDITIONS: Food Insecurity in Post Partum Women
Keywords: Food is Medicine (FIM); food insecurity; free delivered nutritious meals; food boxes; Community Health Workers; The University of Texas Health Science Center at Houston School of Public Health; Austin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- FBM-In person (Experimental)
  Interventions: Other: FBM-In person; Other: home delivered food boxes
- FBM-Virtual (Experimental)
  Interventions: Other: FBM-Virtual; Other: home delivered food boxes
- home delivered food (Active Comparator)
  Interventions: Other: home delivered food boxes

INTERVENTIONS:
Other: FBM-In person — Participants will receive two home visits by a CHW. Each home visit will last about 30 minutes, during which the CHW will assist the woman with community resources and help with enrolling in any state or federal nutrition and medical programs. Furthermore, the participants will be given access to a private Facebook group for nutrition, health education, and social support. Home visits will occur during the second and fifth weeks of the study.
  Arms: FBM-In person
Other: FBM-Virtual — Participants will receive access to a virtual platform which will have information on national, state, and local food and medical resources, as well as local community resources, and will have access to a private Facebook group for nutrition, health education, and social support.
  Arms: FBM-Virtual
Other: home delivered food boxes — Participants will receive weekly deliveries of a box containing fresh produce and staple goods (approximately 5 meals a week), culturally tailored meals (6 meals a week), and prepared fruit, vegetable and grain-forward meal kits (4 units a week) plus standard nutrition education materials consisting of recipes inside of the boxes. Each participant will receive one box for eight consecutive weeks.

SUMMARY:
The purpose of this study is to compare the short-term and long term impacts of Food is the Best Medicine (FBM)-Virtual on diet quality, food security status, breastfeeding rates, mental health status, rates of home cooking, and rationing coping strategies relative to FBM-In Person among food insecure, postpartum women and to compare implementation outcomes across the FBM-Virtual and FBM-In Person using process data collected from the participants, Community Health Worker (CHW)s, and partner organizations.

ELIGIBILITY:
Inclusion Criteria:

* food insecure
* to communicate in English or Spanish.

Exclusion Criteria:

* not living within the food produce zip code delivery radius
* having any dietary allergies.

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 100 (Estimated)
Dates: Start 2024-01-01 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2025-06-30 (Estimated)

PRIMARY OUTCOMES:
Change in level of household food insecurity experienced as assessed by the US Household Food Security questionnaire | Baseline, immediately after intervention (within 2 weeks of completion of intervention), three months after end of intervention
  This is an 6 item questionnaire . Raw score will be reported and score ranges from 0-6. Raw score of 0-1 shows high or marginal food security, raw score of 2- indicates low food security and raw score of 5-6 shows very low food insecurity.
Change in quality of diet as assessed by number of times participants ate certain food items in the past month as reported in the questionnaire | Baseline, immediately after intervention (within 2 weeks of completion of intervention), three months after end of intervention
  This data will be reported categorically for 14 different food items as follows:
  1. fruit
  2. green leafy or lettuce salad
  3. fried potatoes
  4. other kind of potatoes
  5. refired/baked/ cooked beans
  6. other vegetables that were not deep-fried
  7. salsa made with tomato
  8. pizza
  9. tomato sauce
  10. lean protein
  11. plant-based protein
  12. brown rice or other cooked whole grains
  13. whole grain bread
  14. regular soda/pop
Number of participants that initiated breastfeeding as assessed by the pre test questionnaire | Baseline
Total duration of breastfeeding time as assessed by the post test questionnaires | end of study (after 8 weeks of food delivery boxes)
Total duration of breastfeeding time as assessed by the post test questionnaires | 3 months follow up
Change in number of participants who showed signs of depression as assessed by the Edinburgh Postnatal Depression Scale (EPDS) | Baseline, immediately after intervention (within 2 weeks of completion of intervention), three months after end of intervention
  This is a 10 item questionnaire , range of score for each item is 0-3 for a total score range of 0-30, score above 12 is worse outcome
Change in number of cooked meals as assessed by the number of home cooked meals made from scratch during the past week | Baseline, immediately after intervention (within 2 weeks of completion of intervention), three months after end of intervention
  Participant will be asked how often he/she or anyone else in the family prepared breakfast from scratch during the past week, lunch from scratch during the past week or dinner from scratch during the past week. The responses from the 3 items will be summed to determine the number of home cooked meals during past week.
Change in financial stress as assessed by the financial stress questionnaire | Baseline, immediately after intervention (within 2 weeks of completion of intervention), three months after end of intervention
  Scores for three questions from the Financial Stress Scale will be used and each will be scored from 0(never) to 6(Always) for a score range of 0-18; 18 being highest level of financial stress.
Percentage of participants that face financial challenges as assessed by the Financial Self-Efficacy Scale | Baseline, immediately after intervention (within 2 weeks of completion of intervention), three months after end of intervention
  A single item from the Financial Self Efficacy scale will be used.

CONTACTS AND LOCATIONS:
Overall Officials: Alexandra van den Berg, MPH, PhD, Principal Investigator — The University of Texas Health Science Center, Houston
Locations (2):
- United States (2):
  - Ascension Seton Medical Center, Austin, Texas
  - The University of Texas Health Science Center at Houston, Houston, Texas

IPD SHARING:
Plan to Share IPD: No